CLINICAL TRIAL: NCT00094653
Title: A Randomized, Double-Blind, Multicenter Study Comparing MDX-010 Monotherapy, MDX-010 in Combination With a Melanoma Peptide Vaccine, and Melanoma Vaccine Monotherapy in HLA-A2*0201-Positive Patients With Previously Treated Unresectable Stage III or IV Melanoma
Brief Title: MDX-010 Antibody, MDX-1379 Melanoma Vaccine, or MDX-010/MDX-1379 Combination Treatment for Patients With Unresectable or Metastatic Melanoma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Study Director, Bristol-Myers Squibb
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MDX010-20; CA184-002 (Other: BMS)
Record Dates: First submitted 2004-10-21; First posted 2004-10-22 (Estimated); Results first posted 2011-06-23 (Estimated); Last update posted 2011-07-11 (Estimated); Status verified 2011-06

CONDITIONS: Melanoma; Metastases
Keywords: melanoma; metastatic melanoma; skin cancer
MeSH Terms: conditions — Melanoma; Neoplasm Metastasis; Skin Neoplasms | interventions — Ipilimumab; Antibodies, Monoclonal; gp100 Melanoma Antigen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Active Comparator): Melanoma Peptide Vaccine (MDX-1379) (gp100) + Placebo
  Interventions: Biological: MDX-1379 (gp100) Melanoma Peptide Vaccine
- 2 (Experimental): MDX-010 (ipilimumab) + MDX-1379 (gp100) (Melanoma Peptide Vaccine)
  Interventions: Drug: MDX-010 (anti-CTLA4) monoclonal antibody; Biological: MDX-1379 (gp100) Melanoma Peptide Vaccine
- 3 (Active Comparator): MDX-010 (ipilimumab) + Placebo
  Interventions: Drug: MDX-010 (anti-CTLA4) monoclonal antibody

INTERVENTIONS:
Drug: MDX-010 (anti-CTLA4) monoclonal antibody — 3mg/kg (intravenous [iv] infusion over 90 minutes), every 3 weeks for 4 doses
  Other Names: ipilimumab
  Arms: 2; 3
Biological: MDX-1379 (gp100) Melanoma Peptide Vaccine — 2mL (2 subcutaneous injections of 2 mL each, 1 to each thigh), every 3 weeks for 4 doses.
  Other Names: melanoma peptide vaccine
  Arms: 1; 2

SUMMARY:
The purpose of this study is to determine the safety and efficacy of MDX-010 (ipilimumab, BMS-734016) (anti-CTLA4) in combination with MDX-1379 (gp100, BMS-734019) in patients with previously treated, unresectable Stage III or IV melanoma. Survival time will be evaluated, as well as patient responses and time to disease progression. Eligible patients are those who in response to a single regimen containing interleukin-2 (IL-2), dacarbazine, and/or temozolomide, have 1) relapsed following an objective response (partial response/complete response [PR/CR]); 2) failed to demonstrate an objective response (PR/CR); or 3) could not tolerate such a regimen due to unacceptable toxicity. Patients will be randomized into one of three groups, and will receive one of the following treatments: MDX-010 alone, MDX-1379 alone, or MDX-010 in combination with MDX-1379.

DETAILED DESCRIPTION:
Melanoma accounts for approximately 5% of all skin cancers in the United States, but it accounts for about 75% of all skin cancer deaths. In 2004, the expected prevalence of melanoma is 627,252, with about 119,178 of these cases being Stage III or IV (metastatic melanoma). First line treatments for metastatic melanoma, usually IL-2, dacarbazine and/or temozolomide, are associated with significant toxicities. MDX-010 (anti-CTLA4) antibodies are designed to keep the immune system running by blocking CTLA-4 from down-regulating T cell activation. MDX-1379 is made up of two peptides that are pieces of a bigger melanoma protein (gp100). These peptides bind to HLA-A2 which is then recognized by T cells.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with malignant melanoma
* Measurable unresectable Stage III or IV melanoma
* HLA-A*0201 positive
* Previous treatment with & failure/relapse/inability to tolerate IL-2, dacarbazine and/or temozolomide
* At least 4 weeks since prior treatment
* Negative pregnancy
* Life expectancy greater than 4 months
* Eastern Cooperative Oncology Group (ECOG) performance of 0 or 1
* Required lab values
* Human Immunodeficiency Virus (HIV), Hepatitis B Virus (HBV), Hepatitis C Virus (HCV) negative

Exclusion Criteria:

* Prior malignancies which the patient has not been disease free for over 5 years, except treated and cured basal or squamous cell skin cancer, superficial bladder cancer, carcinoma in situ of the cervix, or any other cancer
* Ocular melanoma
* Active, untreated central nervous system (CNS) metastasis
* Prior treatment with MDX-010 (anti-CTLA4) antibody
* Prior treatment with any cancer therapeutic vaccine
* Active autoimmune disease or history of autoimmune disease
* Pregnancy or nursing
* Hypersensitivity to Incomplete Freund's Adjuvant (IFA) (Montanide ISA-51)
* Underlying medical conditions deemed hazardous if treated with study drug
* Concomitant therapy with anti-melanoma drugs, chemotherapies, other investigational therapies, chronic use of systemic corticosteroids
* Unable to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1783 (Actual)
Dates: Start 2004-09; Primary Completion 2009-08 (Actual); Study Completion 2009-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (208):
- United States (109):
  - Arizona Cancer Center, Tucson, Arizona
  - University Medical Center, Tucson, Arizona
  - City of Hope National Medical Center, Duarte, California
  - San Diego Cancer Center, Encinitas, California
  - La Jolla Hematology and Oncology Medical Group, La Jolla, California
  - Scripps Cancer Center, La Jolla, California
  - Moores UCSD Cancer Center, La Jolla, California
  - Pacific Shores Medical Group, Long Beach, California
  - Cancer Institute Medical Group, Inc, Los Angeles, California
  - The Angeles Clinic and Research Institute, Los Angeles, California
  - USC/Norris Comprehensive Cancer Center, Los Angeles, California
  - North County Oncology Medical Clinical, Inc., Oceanside, California
  - City of Hope Medical Group, Pasadena, California
  - University of California, San Diego, San Diego, California
  - St. Mary's Medical Center - Northern California Melanoma Center, San Francisco, California
  - Cancer Institute Medical Group, Inc, Santa Monica, California
  - San Diego Cancer Center, Vista, California
  - Anschutz Cancer Pavilion, Aurora, Colorado
  - Rocky Mountain Cancer Centers, Aurora, Colorado
  - University of Colorado Health Sciences Center, Aurora, Colorado
  - Rocky Mountain Cancer Centers, Boulder, Colorado
  - Rocky Mountain Cancer Centers, Colorado Springs, Colorado
  - Rocky Mountain Cancer Centers, Denver, Colorado
  - University of Colorado Hospital, Denver, Colorado
  - Rocky Mountain Cancer Centers, Lakewood, Colorado
  - Rocky Mountain Cancer Centers, Littleton, Colorado
  - Rocky Mountain Cancer Centers, Lone Tree, Colorado
  - Rocky Mountain Cancer Centers, Longmont, Colorado
  - Yale University School of Medicine - Oncology Outpatient Clinic, New Haven, Connecticut
  - Mount Sinai Comprehensive Cancer Center at Aventura, Aventura, Florida
  - Memorial Regional Cancer Center, Hollywood, Florida
  - Shands Jacksonville, Jacksonville, Florida
  - University of Florida/Jacksonville Faculty Clinic, Jacksonville, Florida
  - Jackson Memorial Hospital & Clinics, Miami, Florida
  - University of Miami Hospital & Clinics, Miami, Florida
  - Mount Sinai Comprehensive Cancer Center, Miami Beach, Florida
  - Mount Sinai Medical Center, Miami Beach, Florida
  - M.D. Anderson Cancer Center Orlando, Orlando, Florida
  - Palm Beach Cancer Institute, Palm Beach Gardens, Florida
  - H. Lee Moffitt Cancer Center & Research Institute, Tampa, Florida
  - Palm Beach Cancer Institute, Wellington, Florida
  - Palm Beach Cancer Institute, West Palm Beach, Florida
  - Emory University Hospital-Winship Cancer Institute, Atlanta, Georgia
  - Cancer Care Specialists of Central IL, Decatur, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Cancer Care Specialists of Central IL, Effingham, Illinois
  - Cardinal Bernardin Cancer Center, Loyola Unv. Med. Ctr., Maywood, Illinois
  - Center for Cancer Care at Goshen Health System, Goshen, Indiana
  - Indiana Oncology Hematology Consultants North, Indianapolis, Indiana
  - American Health Network of IN, LLC, Indianapolis, Indiana
  - Indiana Oncology Hematology South, Indianapolis, Indiana
  - Indiana Oncology Hematology Consutants of Noblesville, Noblesville, Indiana
  - Central Baptist Hospital, Lexington, Kentucky
  - James Graham Brown Cancer Center, Louisville, Kentucky
  - Norton Hospital, Louisville, Kentucky
  - University of Louisville Hospital, Louisville, Kentucky
  - Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland
  - Franklin Square Hospital Center, Baltimore, Maryland
  - Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Lutherville, Maryland
  - Beth Isreal Dec Medical Center, Boston, Massachusetts
  - Brigham and Womens Hospital, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Henry Ford Medical Center, Dearborn, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - Henry Ford Medical Center- West Bloomfield, West Bloomfield, Michigan
  - Humphrey Cancer Center, Coon Rapids, Minnesota
  - Humphrey Cancer Center, Fridley, Minnesota
  - Hubert H Humphrey Cancer Center, Robbinsdale, Minnesota
  - Family Cancer Center, Olive Branch, Mississippi
  - Ellis Fischel Cancer Center, Columbia, Missouri
  - St. Joseph Oncology, Inc, Saint Joseph, Missouri
  - Barnes Jewish Hospital, St Louis, Missouri
  - Washington Unv. School of Med./ Siteman Cancer Center, St Louis, Missouri
  - Hackensack University Medical Center, Hackensack, New Jersey
  - The Cancer Center at Hackensack University Medical Center, Hackensack, New Jersey
  - Hematology-Oncology Associates of Northern NJ, PA, Morristown, New Jersey
  - Robert Wood Johnson University Hospital, New Brunswick, New Jersey
  - The Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Overlook Oncology Center, Summit, New Jersey
  - New Mexico Oncology Hematology Consultants, Ltd., Albuquerque, New Mexico
  - Hematology-Oncology Associates of CNY, East Syracuse, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Columbia University Medical Center, Irving Center for Clinical Research, New York, New York
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - The Christ Hospital Cancer Center, Cincinnati, Ohio
  - The Cleveland Clinic Foundation, Cleveland, Ohio
  - Providence Portland Medical Center, Portland, Oregon
  - The Oregon Clinical, Portland, Oregon
  - Penn State Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Thomas Jefferson University Hosptital, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Hillman Cancer Research Pavilion, Pittsburgh, Pennsylvania
  - Hillman Cancer Center, Pittsburgh, Pennsylvania
  - University of Pittsburgh Cancer Institute, Pittsburgh, Pennsylvania
  - Cancer Centers of the Carolinas, Easley, South Carolina
  - Cancer Centers of the Carolinas, Greenville, South Carolina
  - Cancer Centers of the Carolinas, Seneca, South Carolina
  - Cancer Centers of the Carolinas, Spartanburg, South Carolina
  - Family Cancer Center, Bartlett, Tennessee
  - Family Cancer Center, Collierville, Tennessee
  - Family Cancer Center, Memphis, Tennessee
  - The West Clinic, Memphis, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Arlington Cancer Center, Arlington, Texas
  - Center for Oncology Research and Treatment, Dallas, Texas
  - Joe Arrington Cancer Research and Treatment Center, Lubbock, Texas
  - Center for Oncology Research and Treatment, Richardson, Texas
  - Huntsman Cancer Institute, Salt Lake City, Utah
  - Fletcher Allen Health Care, Burlington, Vermont
- Argentina (14):
  - Hospital Municipal de Oncoligia Maria Curie, Ciudad de Buenos Aires, Buenos Aires
  - Instituto Medico Platense, La Plata, Buenos Aires
  - ISIS Clinica Especializada, Santa Fe, Santa Fe Province
  - Hospital Militar Central, Buenos Aires
  - Instituto Medico Especializado Alexander Fleming, Buenos Aires
  - Hospital Britanico de Buenos Aires, Ciudad de Buenos Aires
  - Hospital Municipal de Oncologia Maria Curie, Ciudad de Buenos Aires
  - Hospital General de Agudos Carlos G. Durand, Ciudad de Buenos Aires
  - Instituto de Oncologia Angel H. Roffo, Ciudad de Buenos Aires
  - Hospital Militar Central, Ciudad de Buenos Aires
  - Instituto Alexander Fleming, Ciudad de Buenos Aires
  - Hospital Privado de Cordoba S.A., Córdoba
  - Hospital Privado Centro Medico de Cordoba S.A., Córdoba
  - ISIS Clinica Especializada, Santa Fe
- Belgium (6):
  - Institut Jules Bordet, Brussels
  - Erasme Hospital, Free Universtiy of Brussels, Brussels
  - Erasme Hospital, Brussels
  - U.Z. Gent, Ghent
  - Universitair Ziekenhuis Gasthuisberg, Leuven
  - Cliniques Universitaires UCL de Mont-Godinne, Yvoir
- Brazil (17):
  - Hospital Araujo Jorge da Associacoa de Combate ao Cancer em Goias, Goiânia, Goiás
  - Pro Onco Centro Tratamento Oncologico, Londrina, Paraná
  - Hospital Sao Lucas da PUCRS, Porto Alegre, Rio Grande do Sul
  - Fundacao Pio XII - Hospital de Cancer de Barretos, Barretos, São Paulo
  - Fundacoa Hospital Amaral Carvalho, Jaú, São Paulo
  - Santo Andre Diagnosticos aTratamentos, Santo André, São Paulo
  - Sociedade Beneficante de Sennores - Hospital Sino Libante, São Paulo, São Paulo
  - Hospital de Cancer de Barretos - Fundacao Pio XII, Barretos - SP
  - Biocor - Hosp. de Doencas Cardiovasculares Ltda., Belo Horizonte - MG
  - Hospital Araujo Jorge, Goiania - GO
  - Pro Onco Centro Tratemento Oncologico, Londrina - PR
  - Fundacao Central Sul-Americana para o Desenvolvimento de Drogas Anticancer-SOAD, Porto Alegre
  - Fund. SOAD / HC de Porto Alegre, Porto Alegre - RS
  - Hospital Sao Lucas - PUCRS, Porto Alegre - RS
  - Santo Andre Diagnosticos e Tratamentos Ltda., Santo Andre-SP
  - HC-FMUSP, Sao Paulo - SP
  - Hospital Sirio Labanes, Sao Paulo-SP
- Canada (9):
  - Tom Baker Cancer Centre, Calgary, Alberta
  - Cross Cancer Institute, Edmonton, Alberta
  - CancerCare Manitoba, Winnipeg, Manitoba
  - Dr. H. Bliss Murphy Cancer Centre, St. John's, Newfoundland and Labrador
  - Cancer Centre of Southeastern Ontario at KGH, Kingston, Ontario
  - London Regional Cancer Program, London, Ontario
  - The Ottawa Hospital Regional Cancer Centre, Ottawa, Ontario
  - Princess Margaret Hospital, Toronto, Ontario
  - Sir Mortimer B. Davis - Jewish General Hospital, Montreal, Quebec
- Chile (5):
  - Instituto Nacional del Cancer, Independencia, Santiago Metropolitan
  - Clinica Davila, Recoleta, Santiago Metropolitan
  - Fundacion Arturo Lopez Perez, Santiago, Santiago Metropolitan
  - Hospital Barros Luco, Santiago, Santiago Metropolitan
  - Clinica Renaca, Reñaca, Vina Del Mar
- France (11):
  - Centre Oscar Lambret, Lille
  - Centre Leon Berard, Lyon
  - Hopital Sainte-Marguerite, Marseille
  - Hopital Saint-Eloi, Montpellier
  - Hotel Dieu, Nantes
  - Centre Antoine Lacassagne, Nice
  - Hopital Saint-Louis, Paris
  - Centre Eugene Marquis, Rennes
  - Centre-Hospitalier Universitaire de Saint-Etienne, Saint-Etienne
  - Centre Alexis Vautrin, Vandœuvre-lès-Nancy
  - Institut Gustave Roussy (IGR), Villejuif
- Germany (14):
  - Klinik fur und Poliklinik fur Dermatologie, Venerologie und Allergologie, Hufelandstr. 55, Hesse
  - Klinikum Augsburg, Augsburg
  - Charite Universitaets medizin Berlin, Berlin
  - Charite-Universitaetsmedizin Berlin, Campus Benjamin Franklin, Berlin
  - Universitaetsklinikum Dusseldorf, Düsseldorf
  - Universitaetsklinikum Erlangen, Erlangen
  - Universitaetsklinikum Essen, Essen
  - Universitaetsklinikum Heidelberg, Heidelberg
  - Klinikum der Friedrich-Schiller-Universitaet Jena, Jena
  - Klinikum Mannheim gGmbH, Mannheim
  - University of Mannheim, Mannheim
  - Klinikum Rechts der Isar / TU Muenchen, München
  - Universitaetsklinikum Tuebingen, Tübingen
  - Universitaetsklinikum Wuerzburg, Würzburg
- Hungary (4):
  - National Institute of Oncology, Budapest
  - University of Debrecen, Medical and Health Sciences Center, Debrecen
  - Semmelweis Hospital, Miskolc
  - University of Szeged, Albert Szent-Gyorgyi Medical and Pharmaceutical Center, Szeged
- Netherlands (3):
  - Antoni Van Leeuwenhoek Ziekenhuis, Amsterdam
  - Vrije Universiteit Medisch Centrum (VUMC), Amsterdam
  - Academisch Ziekenhuis Maastricht, Maastricht
- South Africa (4):
  - Mary Potter Oncology Centre, Groenkloof
  - GVI Oncology, Panorama
  - Mary Potter Oncology Centre, Pretoria
  - Sandton Onocology Medical Research, Sandton
- Switzerland (3):
  - Centre Hospitalier Universitaire Vaudois - CHUV, Lausanne, Rue Du Bugnon 46
  - Centre Hospitalier Universitaire Vaudois - CHUV, Lausanne
  - Dermatologische Klinik Universitatsspital Zurich, Zurich
- United Kingdom (9):
  - St. Luke's Cancer Center, The Royal Surrey County Hospital, Guildford, Surry
  - Velindre Hospital, Cardiff
  - Ninewells Hospital, Dundee
  - Christie Hospital, Manchester
  - Nottingham City Hospital, Nottingham
  - Churchill Hospital, Oxford
  - Poole Hospital, Poole
  - Weston Park Hospital, Sheffield
  - Southampton General, Southampton

REFERENCES:
- [Derived] Larkin J, Hatswell AJ, Nathan P, Lebmeier M, Lee D. The Predicted Impact of Ipilimumab Usage on Survival in Previously Treated Advanced or Metastatic Melanoma in the UK. PLoS One. 2015 Dec 23;10(12):e0145524. doi: 10.1371/journal.pone.0145524. eCollection 2015. PMID 26700304
- [Derived] Koguchi Y, Hoen HM, Bambina SA, Rynning MD, Fuerstenberg RK, Curti BD, Urba WJ, Milburn C, Bahjat FR, Korman AJ, Bahjat KS. Serum Immunoregulatory Proteins as Predictors of Overall Survival of Metastatic Melanoma Patients Treated with Ipilimumab. Cancer Res. 2015 Dec 1;75(23):5084-92. doi: 10.1158/0008-5472.CAN-15-2303. PMID 26627641
- [Derived] Schadendorf D, Hodi FS, Robert C, Weber JS, Margolin K, Hamid O, Patt D, Chen TT, Berman DM, Wolchok JD. Pooled Analysis of Long-Term Survival Data From Phase II and Phase III Trials of Ipilimumab in Unresectable or Metastatic Melanoma. J Clin Oncol. 2015 Jun 10;33(17):1889-94. doi: 10.1200/JCO.2014.56.2736. Epub 2015 Feb 9. PMID 25667295
- [Derived] Johnson DB, Friedman DL, Berry E, Decker I, Ye F, Zhao S, Morgans AK, Puzanov I, Sosman JA, Lovly CM. Survivorship in Immune Therapy: Assessing Chronic Immune Toxicities, Health Outcomes, and Functional Status among Long-term Ipilimumab Survivors at a Single Referral Center. Cancer Immunol Res. 2015 May;3(5):464-9. doi: 10.1158/2326-6066.CIR-14-0217. Epub 2015 Feb 3. PMID 25649350
- [Derived] Hatswell AJ, Pennington B, Pericleous L, Rowen D, Lebmeier M, Lee D. Patient-reported utilities in advanced or metastatic melanoma, including analysis of utilities by time to death. Health Qual Life Outcomes. 2014 Sep 10;12:140. doi: 10.1186/s12955-014-0140-1. PMID 25214238
- [Derived] McDermott D, Haanen J, Chen TT, Lorigan P, O'Day S; MDX010-20 investigators. Efficacy and safety of ipilimumab in metastatic melanoma patients surviving more than 2 years following treatment in a phase III trial (MDX010-20). Ann Oncol. 2013 Oct;24(10):2694-2698. doi: 10.1093/annonc/mdt291. Epub 2013 Aug 13. PMID 23942774
- [Derived] Robert C, Schadendorf D, Messina M, Hodi FS, O'Day S; MDX010-20 investigators. Efficacy and safety of retreatment with ipilimumab in patients with pretreated advanced melanoma who progressed after initially achieving disease control. Clin Cancer Res. 2013 Apr 15;19(8):2232-9. doi: 10.1158/1078-0432.CCR-12-3080. Epub 2013 Feb 26. PMID 23444228
- [Derived] Weber JS, Dummer R, de Pril V, Lebbe C, Hodi FS; MDX010-20 Investigators. Patterns of onset and resolution of immune-related adverse events of special interest with ipilimumab: detailed safety analysis from a phase 3 trial in patients with advanced melanoma. Cancer. 2013 May 1;119(9):1675-82. doi: 10.1002/cncr.27969. Epub 2013 Feb 7. PMID 23400564
- [Derived] Revicki DA, van den Eertwegh AJ, Lorigan P, Lebbe C, Linette G, Ottensmeier CH, Safikhani S, Messina M, Hoos A, Wagner S, Kotapati S. Health related quality of life outcomes for unresectable stage III or IV melanoma patients receiving ipilimumab treatment. Health Qual Life Outcomes. 2012 Jun 13;10:66. doi: 10.1186/1477-7525-10-66. PMID 22694829
- [Derived] Hodi FS, O'Day SJ, McDermott DF, Weber RW, Sosman JA, Haanen JB, Gonzalez R, Robert C, Schadendorf D, Hassel JC, Akerley W, van den Eertwegh AJ, Lutzky J, Lorigan P, Vaubel JM, Linette GP, Hogg D, Ottensmeier CH, Lebbe C, Peschel C, Quirt I, Clark JI, Wolchok JD, Weber JS, Tian J, Yellin MJ, Nichol GM, Hoos A, Urba WJ. Improved survival with ipilimumab in patients with metastatic melanoma. N Engl J Med. 2010 Aug 19;363(8):711-23. doi: 10.1056/NEJMoa1003466. Epub 2010 Jun 5. PMID 20525992

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of the 1783 participants who enrolled and were screened for study participation, a total of 676 subjects were randomized.
Groups:
- Ipilimumab Plus gp100: Ipilimumab was administered at a dosage of 3 mg/kg as an intravenous (IV) infusion administered over 90 minutes every 3 weeks for a total of 4 doses, together with gp100. Gp100 consisted of 2 separate peptide components: Peptide A, a peptide with sequence YLEPGPVTV (gp100:280-288[288V]) and Peptide B, a peptide with the sequence IMDQVPFSV (gp100:209-217[210M]). Each peptide was prepared with Montanide ISA-51. One dose of gp100 consisted of the administration of Peptide A, at a dosage of 2 mL or 1 mg, and Peptide B, at a dosage of 2 mL or 1 mg. After Week 12, subjects who met re-induction criteria could receive further cycles of their randomized study therapy.
- Ipilimumab Monotherapy: Ipilimumab was administered at a dosage of 3 mg/kg as an intravenous (IV) infusion administered over 90 minutes every 3 weeks for a total of 4 doses, together with matching vaccine placebo. The vaccine placebo consisted of sterile 0.9% sodium chloride. After Week 12, subjects who met re-induction criteria could receive further cycles of their randomized study therapy.
- gp100: Gp100 consisted of 2 separate peptide components: Peptide A, a peptide with sequence YLEPGPVTV (gp100:280-288[288V]) and Peptide B, a peptide with the sequence IMDQVPFSV (gp100:209-217[210M]). Each peptide was prepared with Montanide ISA-51. One dose of gp100 consisted of the administration of Peptide A, at a dosage of 2 mL or 1 mg, and Peptide B, at a dosage of 2 mL or 1 mg. After Week 12, subjects who met re-induction criteria could receive further cycles of their randomized study therapy.
Period: Overall Study
Arm/Group | Ipilimumab Plus gp100 | Ipilimumab Monotherapy | gp100
Started | 403 | 137 | 136
Treated | 381 | 131 | 131
Completed | 82 | 31 | 10
Not Completed | 321 | 106 | 126
Not completed — Death | 306 | 100 | 119
Not completed — Subject Withdrew Consent | 10 | 2 | 3
Not completed — Other | 2 | 2 | 2
Not completed — Lost to Follow-up | 3 | 2 | 1
Not completed — Protocol Violation | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ipilimumab Plus gp100 | Ipilimumab Monotherapy | gp100 | Total
Number analyzed (Participants) | 403 | 137 | 136 | 676
Age Continuous [Mean (Full Range); unit: years] | 55.6 [24 to 84] | 56.8 [19 to 88] | 57.4 [23 to 90] | 56.2 [19 to 90]
Age, Customized [Number; unit: participants]
  < 65 years | 291 | 95 | 94 | 480
  >=65 years | 112 | 42 | 42 | 196
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 156 | 56 | 63 | 275
  Male | 247 | 81 | 73 | 401
Race/Ethnicity, Customized [Number; unit: Participants]
  White | 380 | 129 | 129 | 638
  Black | 3 | 1 | 1 | 5
  Hispanic | 18 | 7 | 5 | 30
  Other | 2 | 0 | 1 | 3
Duration of Melanoma [Mean (Full Range); unit: years] — Duration of melanoma is the number of years from date of initial diagnosis to the date of randomization. The randomization of 1 participant in the ipilumumab monotherapy cohort was prior to the initial diagnostic date. Data for 2 participants in the ipilimumab + gp100 cohort were missing.
  years | 5.09 [0.2 to 38.9] | 4.34 [-0.0 to 35.9] | 5.65 [0.3 to 31.2] | 5.05 [-0.0 to 38.9]
Melanoma Stage [Number; unit: Participants] — The "M" in the TNM (tumor, node, metastasis) system refers to distant metastases-whether, and how far, the cancer has spread outside the original site. M0: There is no evidence that the cancer has spread beyond the original site. M1: The cancer has spread beyond the original site. M1a: The cancer has spread to other areas of skin, underneath the epidermis to the dermis (subcutaneous), or to lymph node(s). M1b: The cancer has spread to the lung(s) only. M1c: The cancer has spread to other organs and/or locations in the body with or without elevated LDH.
  Participants
    M0 | 5 | 1 | 4 | 10
    M1a | 37 | 14 | 11 | 62
    M1b | 76 | 22 | 23 | 121
    M1c | 285 | 100 | 98 | 483
Prior Interleukin-2 Therapy [Number; unit: Participants]
  No | 314 | 105 | 103 | 522
  Yes | 89 | 32 | 33 | 154
Lactate Dehydrogenase [Number; unit: Participants] — Upper limit of normal (ULN) was 250 U/L for most assessments (some variation caused by tests performed at local laboratories).
  Participants
    >upper limit of normal (ULN) | 149 | 53 | 52 | 254
    <=ULN | 252 | 84 | 81 | 417
    unknown | 2 | 0 | 3 | 5

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival (OS) (Time-to-Death) Difference Between MDX-010 in Combination With gp 100 Melanoma Peptide Vaccine Versus gp 100 Melanoma Peptide Vaccine Alone
Description: OS was defined as the time from randomization until death from any cause. If a participant did not expire, the subject was censored at the time of last contact (last known alive date). 95% confidence intervals (CI) for median were computed using Brookmeyer and Crowley method.
Time Frame: From randomization until the end of the study, which was defined as the time at which 481 deaths were observed (264 weeks)
Population: Intent-to-treat population, as randomized. All subjects who were randomized to any treatment group in the study.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Ipilimumab Plus gp100 | gp100
Number analyzed (Participants) | 403 | 136
months | 9.95 [8.48 to 11.50] | 6.44 [5.49 to 8.71]
Statistical Analysis 1: Comparison: Ipilimumab Plus gp100 vs gp100; Test type: Superiority or Other; p = 0.0004, Stratified Log Rank; Hazard Ratio (HR) = 0.68, 95% CI 2-sided [0.55 to 0.85] — Cox model for Hazard ratios (HR) and log-rank test p-values were stratified by baseline M-stage at randomization (M0, M1a, M1b vs. M1c) and prior treatment with IL-2 (Yes vs. No)

2. Secondary Outcome: Overall Survival (OS) (Time-to-Death) Difference Between MDX-010 Monotherapy Versus gp100 Melanoma Peptide Vaccine Alone and MDX-010 in Combination With gp100 Melanoma Peptide Vaccine Versus MDX-010 Monotherapy
Description: as for outcome 1
Time Frame: as for outcome 1
Population: Intent-to-treat population, as randomized. All subjects who were randomized to any treatment group in the study.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Ipilimumab Plus gp100 | Ipilimumab Monotherapy | gp100
Number analyzed (Participants) | 403 | 137 | 136
months | 9.95 [8.48 to 11.50] | 10.12 [8.02 to 13.80] | 6.44 [5.49 to 8.71]
Statistical Analysis 1: Comparison: Ipilimumab Monotherapy vs gp100; Test type: Superiority or Other; p = 0.0026, Stratified Log Rank; Hazard Ratio (HR) = 0.66, 95% CI 2-sided [0.51 to 0.87] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Ipilimumab Plus gp100 vs Ipilimumab Monotherapy; Test type: Superiority or Other; p = 0.7575, Stratified Log Rank; Hazard Ratio (HR) = 1.04, 95% CI 2-sided [0.83 to 1.30] — [estimate comment as in outcome 1, analysis 1]

3. Secondary Outcome: 12-, 18-, and 24-Month Survival Rates
Description: The probability that a subject is alive at 12 months, 18 months, and 24 months following randomization, estimated via the non-parametric method (Kaplan-Meier method). For calculating 95% CI, bootstrap method was used with 20000 simulated trials.
Time Frame: Month 12, Month 18, Month 24
Population: Intent-to-treat population, as randomized. All subjects who were randomized to any treatment group in the study.
Measure: Number (95% Confidence Interval); unit: probability
Arm/Group | Ipilimumab Plus gp100 | Ipilimumab Monotherapy | gp100
Number analyzed (Participants) | 403 | 137 | 136
probability
  12-Month Survival Rate | 0.436 [0.386 to 0.485] | 0.456 [0.370 to 0.541] | 0.253 [0.181 to 0.329]
  18-Month Survival Rate | 0.300 [0.254 to 0.347] | 0.332 [0.249 to 0.417] | 0.163 [0.101 to 0.230]
  24-Month Survival Rate | 0.216 [0.172 to 0.261] | 0.235 [0.160 to 0.315] | 0.137 [0.080 to 0.200]

4. Secondary Outcome: Progression Free Survival (PFS)
Description: PFS was defined as the number of days between the date of randomization and the date of the progression or the date of death. A subject who died without prior progression was considered to have progressed on the date of death. PFS was determined by investigator. 95% confidence intervals (CI) for median were computed using Brookmeyer and Crowley method.
Time Frame: as for outcome 1
Population: Intent-to-treat population, as randomized. All subjects who were randomized to any treatment group in the study. Subjects who neither progressed nor died were censored at the date of the last tumor assessment.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Ipilimumab Plus gp100 | Ipilimumab Monotherapy | gp100
Number analyzed (Participants) | 403 | 137 | 136
months | 2.76 [2.73 to 2.79] | 2.86 [2.76 to 3.02] | 2.76 [2.73 to 2.83]
Statistical Analysis 1: Comparison: Ipilimumab Plus gp100 vs gp100; Test type: Superiority or Other; Hazard Ratio (HR) = 0.81, 95% CI 2-sided [0.66 to 1.00] — Cox model for Hazard ratios (HR) were stratified by M-stage at randomization (M0, M1a, M1b vs. M1c) and prior treatment with IL-2 (Yes vs. No)
Statistical Analysis 2: Comparison: Ipilimumab Monotherapy vs gp100; Test type: Superiority or Other; Hazard Ratio (HR) = 0.64, 95% CI 2-sided [0.50 to 0.83] — [estimate comment as in outcome 4, analysis 1]
Statistical Analysis 3: Comparison: Ipilimumab Plus gp100 vs Ipilimumab Monotherapy; Test type: Superiority or Other; Hazard Ratio (HR) = 1.25, 95% CI 2-sided [1.01 to 1.53] — [estimate comment as in outcome 4, analysis 1]

5. Secondary Outcome: Percentage of Participants With Progression Free Survival (PFS) at Week 12 and Week 24
Description: PFS at Week 12 was defined as the probability that the subject was progression-free at 12 weeks and 24 weeks following the start of randomization. It was computed via Kaplan-Meier method, truncated at Week 12 and Week 24. PFS was determined by investigator. 95% confidence intervals (CI) for median were computed using Brookmeyer and Crowley method.
Time Frame: Week 12, Week 24
Population: Intent-to-treat population, as randomized. All subjects who were randomized to any treatment group in the study.
Measure: Median (95% Confidence Interval); unit: percentage of participants
Arm/Group | Ipilimumab Plus gp100 | Ipilimumab Monotherapy | gp100
Number analyzed (Participants) | 403 | 137 | 136
percentage of participants
  Week 12 | 0.491 [0.441 to 0.539] | 0.577 [0.489 to 0.655] | 0.485 [0.396 to 0.567]
  Week 24 | 0.164 [0.129 to 0.203] | 0.240 [0.171 to 0.315] | 0.100 [0.056 to 0.159]

6. Secondary Outcome: Time to Progression (TTP)
Description: TTP was defined as the number of days between the date of the randomization and date of PD or death due to PD. For subjects who had not progression and remained alive, TTP was censored on the date of last assessment; those who remained alive and had no recorded post-baseline assessment, TTP was censored on the date of randomization; those who remained alive and had randomized but were not treated, TTP was censored at the date of randomization; for those who died without reported disease progression, TTP was censored on the date of death.
Time Frame: from time of randomization to date of PD or death due to PD (end of the study was defined as the time at which 481 deaths were observed [264 weeks])
Population: Intent-to-treat population, as randomized. All subjects who were randomized to any treatment group in the study.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Ipilimumab Plus gp100 | Ipilimumab Monotherapy | gp100
Number analyzed (Participants) | 403 | 137 | 136
months | 2.76 [2.73 to 2.79] | 2.86 [2.76 to 3.02] | 2.76 [2.73 to 2.83]
Statistical Analysis 1: Comparison: Ipilimumab Plus gp100 vs gp100; Test type: Superiority or Other; Hazard Ratio (HR) = 0.81, 95% CI 2-sided [0.66 to 1.00] — [estimate comment as in outcome 4, analysis 1]
Statistical Analysis 2: Comparison: Ipilimumab Monotherapy vs gp100; Test type: Superiority or Other; Hazard Ratio (HR) = 0.64, 95% CI 2-sided [0.50 to 0.83] — [estimate comment as in outcome 4, analysis 1]
Statistical Analysis 3: Comparison: Ipilimumab Plus gp100 vs Ipilimumab Monotherapy; Test type: Superiority or Other; Hazard Ratio (HR) = 1.25, 95% CI 2-sided [1.01 to 1.53] — [estimate comment as in outcome 4, analysis 1]

7. Secondary Outcome: Best Overall Response (BOR): Complete Response (CR), Partial Response (PR), Stable Disease (SD), Progressed Disease (PD)
Description: Investigator's assessment, modified World Health Organization criteria. CR: disappearance of all lesions by 2 consecutive observations >=4 weeks apart, no evidence of PD. PR: >=50% ↓ in sum of products of longest diameter & greatest perpendicular diameter of all target lesions compared to baseline by 2 observations >=4 weeks apart. SD: Neither sufficient ↓ to qualify for PR nor sufficient ↑ to qualify for PD. PD: ↑ >=25% in sum of products of longest diameter & greatest perpendicular diameter of target lesions compared to smallest recorded sum during study, or appearance of >= 1 new lesion.
Time Frame: BOR was determined between Weeks 12 and Week 24 confirmation at least 4 weeks later at Cycle 1.
Population: Intent-to-treat population, as randomized. All subjects who were randomized to any treatment group in the study.
Measure: Number; unit: participants
Arm/Group | Ipilimumab Plus gp100 | Ipilimumab Monotherapy | gp100
Number analyzed (Participants) | 403 | 137 | 136
participants
  Complete Response | 1 | 2 | 0
  Partial Response | 22 | 13 | 2
  Stable Disease | 58 | 24 | 13
  Progressed Disease | 239 | 70 | 89
  Not Evaluated, Missing, or Unknown | 83 | 28 | 32

8. Secondary Outcome: Determination of Best Overall Response Rate (BORR)
Description: Response was based on the investigators' assessment using modified WHO criteria. BORR is defined as the number of subjects whose BOR is complete or partial response (CR or PR) divided by the total number of subjects in the group. BORR was comprised of responder and non-responder. The definition of a responder in BORR was either confirmed CR or PR, and a non-responder was defined as stable disease (SD), progressed disease (PD), unconfirmed CR (uCR), unconfirmed PR (uPR), and not evaluated.
Time Frame: Up to week 24
Population: Intent-to-treat population, as randomized. All subjects who were randomized to any treatment group in the study.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Ipilimumab Plus gp100 | Ipilimumab Monotherapy | gp100
Number analyzed (Participants) | 403 | 137 | 136
percentage of participants | 5.7 [3.7 to 8.4] | 10.9 [6.3 to 17.4] | 1.5 [0.2 to 5.2]
Statistical Analysis 1: Comparison: Ipilimumab Plus gp100 vs gp100; Test type: Superiority or Other; p = 0.0433, Cochran-Mantel-Haenszel — P-values were computed using CMH test stratified by baseline M-stage at randomization (M0, M1a, M1b vs. M1c) and prior IL-2 treatment (Yes vs. No)
Statistical Analysis 2: Comparison: Ipilimumab Monotherapy vs gp100; Test type: Superiority or Other; p = 0.0012, Cochran-Mantel-Haenszel — [p-value comment as in outcome 8, analysis 1]
Statistical Analysis 3: Comparison: Ipilimumab Plus gp100 vs Ipilimumab Monotherapy; Test type: Superiority or Other; p = 0.0402, Cochran-Mantel-Haenszel — [p-value comment as in outcome 8, analysis 1]

9. Secondary Outcome: Time to Response
Description: Time to response was defined as the number of days from the date of randomization to the date when measurement criteria are met for BOR of CR or PR, as determined by investigator.
Time Frame: as for outcome 1
Population: Responder subjects in intent-to-treat population, as randomized. All subjects who were randomized to any treatment group in the study.
Measure: Mean (Full Range); unit: months
Arm/Group | Ipilimumab Plus gp100 | Ipilimumab Monotherapy | gp100
Number analyzed (Participants) | 23 | 15 | 2
months | 3.324 (0.9561) [2.10 to 5.59] | 3.176 (0.7629) [2.60 to 5.52] | 2.743 (0.0697) [2.69 to 2.79]

10. Secondary Outcome: Duration of Response
Description: Kaplan-Meier medians along with Brookmeyer and Crowley 95% confidence intervals (CI) for were computed. Duration of response was defined in subjects whose BOR was CR or PR as the number of days between the date of response (CR or PR) and the date of PD or the date of death (whichever occurs first).
Time Frame: from time of initial drug administration to date of PD or death due to PD (the end of the study was defined as the time at which 481 deaths were observed [264 weeks])
Population: Responders only in intent-to-treat population, as randomized. All subjects who were randomized to any treatment group in the study. Patients who did not progress or died were censored at the date of their last tumor assessment.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Ipilimumab Plus gp100 | Ipilimumab Monotherapy | gp100
Number analyzed (Participants) | 23 | 15 | 2
months | 11.47 [5.36 to NA] — Upper limit of 95% CI was not reached because most subjects were censored and the upper bound was not estimable. | NA [28.09 to NA] — Median duration of response was not reached because of the number of ongoing responses (ie, since most subjects did not progress-die, the median was not reached). | NA [2.00 to NA] — The limited number of responses (2) in the gp100 monotherapy group prevented a median duration from being reached.

11. Secondary Outcome: Disease Control Rate (DCR)
Description: Response was based on the investigators' assessment using modified WHO criteria. DCR is defined as the number of subjects whose BOR is CR, PR, or SD divided by the total number of subjects in the group.
Time Frame: Up to week 24
Population: Intent-to-treat population, as randomized. All subjects who were randomized to any treatment group in the study.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Ipilimumab Plus gp100 | Ipilimumab Monotherapy | gp100
Number analyzed (Participants) | 403 | 137 | 136
percentage of participants | 20.1 [16.3 to 24.3] | 28.5 [21.1 to 36.8] | 11.0 [6.3 to 17.5]
Statistical Analysis 1: Comparison: Ipilimumab Plus gp100 vs gp100; Test type: Superiority or Other; p = 0.0179, Cochran-Mantel-Haenszel — [p-value comment as in outcome 8, analysis 1]
Statistical Analysis 2: Comparison: Ipilimumab Monotherapy vs gp100; Test type: Superiority or Other; p = 0.0002, Cochran-Mantel-Haenszel — [p-value comment as in outcome 8, analysis 1]
Statistical Analysis 3: Comparison: Ipilimumab Plus gp100 vs Ipilimumab Monotherapy; Test type: Superiority or Other; p = 0.0429, Cochran-Mantel-Haenszel — [p-value comment as in outcome 8, analysis 1]

12. Secondary Outcome: Delayed Response (Response Beyond Week 24)
Description: Response was based on the investigators' assessment using modified World Health Organization (WHO) criteria. Delayed response is defined as post Week 24 overall response for the subjects who have PD before or at Week 24. Evaluation of delayed overall response is compared to baseline assessment. Delayed response includes delayed late CR, delayed late PR, delayed late SD, continued PD, unknown, and missing after Week 24. The delayed response of CR and PR also must have been confirmed.
Time Frame: from Week 24 to end of study (the end of the study was defined as the time at which 481 deaths were observed [264 weeks])
Population: Number of subjects with BOR of PR/SD (80 subjects ipi + gp100 , 37 ipi , 15 gp100) plus number of subjects with BOR of PD that had subsequent evaluation (8 ipi + gp100, 3 ipi, 3 gp100).
Measure: Number; unit: participants
Arm/Group | Ipilimumab Plus gp100 | Ipilimumab Monotherapy | gp100
Number analyzed (Participants) | 88 | 40 | 18
participants
  Complete Response Beyond Week 24 | 1 | 3 | 0
  Partial Response Beyond Week 24 | 3 | 2 | 0
  Stable Disease Beyond Week 24 | 3 | 0 | 0

13. Secondary Outcome: Change From Baseline in Health-Related Quality of Life (QOL) as Measured by the European Organization for Research and Treatment of Cancer Core Quality of Life Questionnaire (EORTC QLQ-C30) Instrument at Week 12
Description: The 30 items were grouped into the following: 1 global QOL scale, 5 functional scales (Physical, Role, Cognitive, Emotional, Social), and 9 symptom scales/items (Fatigue, Nausea and Vomiting, Pain, Dyspnea, Sleep Disturbance, Appetite Loss, Constipation, Diarrhea, Financial Impact). All scores were linearly transformed to a 0 to 100 scale. For global QOL and functional items, a higher score represents a better level of functioning (100=best/0=worst). For symptom items, a higher score represents a higher level of symptoms (0=no symptom at all/100=very much severe).
Time Frame: Baseline (Day 1, Cycle1), Week 12
Population: All subjects who received at least 1 dose or any partial dose of study medication. N=number of participants analyzed, n=number of participants with measure at given time points.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Ipilimumab Plus gp100 | Ipilimumab Monotherapy | gp100
Number analyzed (Participants) | 381 | 131 | 131
units on a scale
  Global QOL (n=226, 83, 77) | -7.4 [-10.4 to -4.3] | -8.8 [-13.5 to -4.1] | -10.4 [-15.3 to -5.5]
  Physical (n=226 83, 78) | -6.2 [-8.9 to -3.4] | -5.1 [-9.4 to -0.8] | -10.1 [-14.5 to -5.7]
  Role Change (n=226, 83, 78) | -9.3 [-13.4 to -5.3] | -10.5 [-16.8 to -4.1] | -13.7 [-20.2 to -7.2]
  Cognitive (n=226, 83, 78) | -3.1 [-5.8 to -0.3] | -4.3 [-8.6 to 0.0] | -3.4 [-7.8 to 1.0]
  Emotional (n=227, 83, 78) | -1.5 [-4.2 to 1.1] | -3.6 [-7.7 to 0.6] | -1.5 [-5.8 to 2.7]
  Social (n=227, 83, 76) | -5.6 [-9.2 to -2.0] | -7.5 [-13.2 to -1.9] | -4.2 [-10.1 to 1.8]
  Fatigue (n=226, 82, 78) | 10.6 [7.0 to 14.1] | 12.5 [7.0 to 18.1] | 14.5 [8.8 to 20.2]
  Nausea and Vomiting (n=226, 83, 78) | 4.6 [1.9 to 7.3] | 3.1 [-1.0 to 7.3] | 4.4 [0.1 to 8.7]
  Pain (n=227, 83, 78) | 5.6 [2.0 to 9.3] | 7.9 [2.2 to 13.6] | 11.9 [6.0 to 17.7]
  Dyspnea (n=222, 81, 77) | 3.5 [0.0 to 6.9] | 5.3 [-0.1 to 10.7] | 9.1 [3.6 to 14.6]
  Sleep Disturbance (n=225, 83, 76) | 6.5 [2.3 to 10.7] | 10.1 [3.6 to 16.6] | 11.0 [4.3 to 17.8]
  Appetite Loss (n=225, 83, 78) | 8.5 [4.4 to 12.5] | 11.6 [5.3 to 17.9] | 10.3 [3.8 to 16.8]
  Constipation (n=225, 83, 77) | 5.2 [1.7 to 8.7] | 1.9 [-3.5 to 7.2] | 11.8 [6.2 to 17.4]
  Diarrhea (n=223, 82, 78) | 6.4 [2.8 to 10.1] | 9.1 [3.4 to 14.7] | 2.1 [-3.7 to 7.9]
  Financial Impact (n=226, 83, 76) | 0.0 [-3.2 to 3.2] | 3.1 [-1.9 to 8.1] | 1.7 [-3.5 to 6.9]
Statistical Analysis 1: Comparison: Ipilimumab Plus gp100 vs gp100; Global quality of life change from baseline; Test type: Superiority or Other; p = 0.2805, ANCOVA; Mean Difference (Final Values) = 3.0, 95% CI 2-sided [-2.5 to 8.6] — Least square mean can be defined as a linear combination of estimated effects, from a linear model. These means are based on ANCOVA model with covariate variables as baseline score, M-stage and prior-IL2 treatment at randomization, and treatment
Statistical Analysis 2: Comparison: Ipilimumab Monotherapy vs gp100; Global quality of life change from baseline; Test type: Superiority or Other; p = 0.6300, ANCOVA; Mean Difference (Final Values) = 1.6, 95% CI 2-sided [-5.0 to 8.2] — [estimate comment as in outcome 13, analysis 1]
Statistical Analysis 3: Comparison: Ipilimumab Plus gp100 vs Ipilimumab Monotherapy; Global quality of life change from baseline; Test type: Superiority or Other; p = 0.6026, ANCOVA; Mean Difference (Final Values) = 1.4, 95% CI 2-sided [-3.9 to 6.8] — [estimate comment as in outcome 13, analysis 1]
Statistical Analysis 4: Comparison: Ipilimumab Plus gp100 vs gp100; Physical change from baseline; Test type: Superiority or Other; p = 0.1219, ANCOVA; Mean Difference (Final Values) = 3.9, 95% CI 2-sided [-1.1 to 8.9] — [estimate comment as in outcome 13, analysis 1]
Statistical Analysis 5: Comparison: Ipilimumab Monotherapy vs gp100; Physical change from baseline; Test type: Superiority or Other; p = 0.0978, ANCOVA; Mean Difference (Final Values) = 5.0, 95% CI 2-sided [-0.9 to 11.0] — [estimate comment as in outcome 13, analysis 1]
Statistical Analysis 6: Comparison: Ipilimumab Plus gp100 vs Ipilimumab Monotherapy; Physical change from baseline; Test type: Superiority or Other; p = 0.6590, ANCOVA; Mean Difference (Final Values) = -1.1, 95% CI 2-sided [-6.0 to 3.8] — [estimate comment as in outcome 13, analysis 1]
Statistical Analysis 7: Comparison: Ipilimumab Plus gp100 vs gp100; Role change, change from baseline; Test type: Superiority or Other; p = 0.2480, ANCOVA; Mean Difference (Final Values) = 4.3, 95% CI 2-sided [-3.0 to 11.7] — [estimate comment as in outcome 13, analysis 1]
Statistical Analysis 8: Comparison: Ipilimumab Monotherapy vs gp100; Role change, change from baseline; Test type: Superiority or Other; p = 0.4742, ANCOVA; Mean Difference (Final Values) = 3.2, 95% CI 2-sided [-5.6 to 12.0] — [estimate comment as in outcome 13, analysis 1]
Statistical Analysis 9: Comparison: Ipilimumab Plus gp100 vs Ipilimumab Monotherapy; Role change, change from baseline; Test type: Superiority or Other; p = 0.7597, ANCOVA; Mean Difference (Final Values) = 1.1, 95% CI 2-sided [-6.1 to 8.3] — [estimate comment as in outcome 13, analysis 1]
Statistical Analysis 10: Comparison: Ipilimumab Plus gp100 vs gp100; Cognitive change from baseline; Test type: Superiority or Other; p = 0.9119, ANCOVA; Mean Difference (Final Values) = 0.3, 95% CI 2-sided [-4.7 to 5.2] — [estimate comment as in outcome 13, analysis 1]
Statistical Analysis 11: Comparison: Ipilimumab Monotherapy vs gp100; Cognitive change from baseline; Test type: Superiority or Other; p = 0.7616, ANCOVA; Mean Difference (Final Values) = -0.9, 95% CI 2-sided [-6.9 to 5.0] — [estimate comment as in outcome 13, analysis 1]
Statistical Analysis 12: Comparison: Ipilimumab Plus gp100 vs Ipilimumab Monotherapy; Cognitive change from baseline; Test type: Superiority or Other; p = 0.6266, ANCOVA; Mean Difference (Final Values) = 1.2, 95% CI 2-sided [-3.6 to 6.0] — [estimate comment as in outcome 13, analysis 1]
Statistical Analysis 13: Comparison: Ipilimumab Plus gp100 vs gp100; Emotional change from baseline; Test type: Superiority or Other; p = 0.9984, ANCOVA; Mean Difference (Final Values) = 0.0, 95% CI 2-sided [-4.8 to 4.8] — [estimate comment as in outcome 13, analysis 1]
Statistical Analysis 14: Comparison: Ipilimumab Monotherapy vs gp100; Emotional change from baseline; Test type: Superiority or Other; p = 0.4873, ANCOVA; Mean Difference (Final Values) = -2.0, 95% CI 2-sided [-7.8 to 3.7] — [estimate comment as in outcome 13, analysis 1]
Statistical Analysis 15: Comparison: Ipilimumab Plus gp100 vs Ipilimumab Monotherapy; Emotional change from baseline; Test type: Superiority or Other; p = 0.3938, ANCOVA; Mean Difference (Final Values) = 2.0, 95% CI 2-sided [-2.7 to 6.7] — [estimate comment as in outcome 13, analysis 1]
Statistical Analysis 16: Comparison: Ipilimumab Plus gp100 vs gp100; Social change from baseline; Test type: Superiority or Other; p = 0.6695, ANCOVA; Mean Difference (Final Values) = -1.4, 95% CI 2-sided [-8.1 to 5.2] — [estimate comment as in outcome 13, analysis 1]
Statistical Analysis 17: Comparison: Ipilimumab Monotherapy vs gp100; Social change from baseline; Test type: Superiority or Other; p = 0.4041, ANCOVA; Mean Difference (Final Values) = -3.4, 95% CI 2-sided [-11.3 to 4.6] — [estimate comment as in outcome 13, analysis 1]
Statistical Analysis 18: Comparison: Ipilimumab Plus gp100 vs Ipilimumab Monotherapy; Social change from baseline; Test type: Superiority or Other; p = 0.5538, ANCOVA; Mean Difference (Final Values) = 1.9, 95% CI 2-sided [-4.5 to 8.3] — [estimate comment as in outcome 13, analysis 1]
Statistical Analysis 19: Comparison: Ipilimumab Plus gp100 vs gp100; Fatigue change from baseline; Test type: Superiority or Other; p = 0.2259, ANCOVA; Mean Difference (Final Values) = -3.9, 95% CI 2-sided [-10.3 to 2.4] — [estimate comment as in outcome 13, analysis 1]
Statistical Analysis 20: Comparison: Ipilimumab Monotherapy vs gp100; Fatigue change from baseline; Test type: Superiority or Other; p = 0.6168, ANCOVA; Mean Difference (Final Values) = -2.0, 95% CI 2-sided [-9.6 to 5.7] — [estimate comment as in outcome 13, analysis 1]
Statistical Analysis 21: Comparison: Ipilimumab Plus gp100 vs Ipilimumab Monotherapy; Fatigue change from baseline; Test type: Superiority or Other; p = 0.5329, ANCOVA; Mean Difference (Final Values) = -2.0, 95% CI 2-sided [-8.2 to 4.3] — [estimate comment as in outcome 13, analysis 1]
Statistical Analysis 22: Comparison: Ipilimumab Plus gp100 vs gp100; Nausea and Vomiting change from baseline; Test type: Superiority or Other; p = 0.9397, ANCOVA; Mean Difference (Final Values) = 0.2, 95% CI 2-sided [-4.7 to 5.0] — [estimate comment as in outcome 13, analysis 1]
Statistical Analysis 23: Comparison: Ipilimumab Monotherapy vs gp100; Nausea and Vomiting change from baseline; Test type: Superiority or Other; p = 0.6716, ANCOVA; Mean Difference (Final Values) = -1.3, 95% CI 2-sided [-7.1 to 4.6] — [estimate comment as in outcome 13, analysis 1]
Statistical Analysis 24: Comparison: Ipilimumab Plus gp100 vs Ipilimumab Monotherapy; Nausea and Vomiting change from baseline; Test type: Superiority or Other; p = 0.5497, ANCOVA; Mean Difference (Final Values) = 1.4, 95% CI 2-sided [-3.3 to 6.2] — [estimate comment as in outcome 13, analysis 1]
Statistical Analysis 25: Comparison: Ipilimumab Plus gp100 vs gp100; Pain change from baseline; Test type: Superiority or Other; p = 0.0625, ANCOVA; Mean Difference (Final Values) = -6.3, 95% CI 2-sided [-12.8 to 0.3] — [estimate comment as in outcome 13, analysis 1]
Statistical Analysis 26: Comparison: Ipilimumab Monotherapy vs gp100; Pain change from baseline; Test type: Superiority or Other; p = 0.3214, ANCOVA; Mean Difference (Final Values) = -4.0, 95% CI 2-sided [-11.9 to 3.9] — [estimate comment as in outcome 13, analysis 1]
Statistical Analysis 27: Comparison: Ipilimumab Plus gp100 vs Ipilimumab Monotherapy; Pain change from baseline; Test type: Superiority or Other; p = 0.4898, ANCOVA; Mean Difference (Final Values) = -2.3, 95% CI 2-sided [-8.7 to 4.2] — [estimate comment as in outcome 13, analysis 1]
Statistical Analysis 28: Comparison: Ipilimumab Plus gp100 vs gp100; Dyspnea change from baseline; Test type: Superiority or Other; p = 0.0761, ANCOVA; Mean Difference (Final Values) = -5.6, 95% CI 2-sided [-11.8 to 0.6] — [estimate comment as in outcome 13, analysis 1]
Statistical Analysis 29: Comparison: Ipilimumab Monotherapy vs gp100; Dyspnea change from baseline; Test type: Superiority or Other; p = 0.3187, ANCOVA; Mean Difference (Final Values) = -3.8, 95% CI 2-sided [-11.2 to 3.7] — [estimate comment as in outcome 13, analysis 1]
Statistical Analysis 30: Comparison: Ipilimumab Plus gp100 vs Ipilimumab Monotherapy; Dyspnea change from baseline; Test type: Superiority or Other; p = 0.5548, ANCOVA; Mean Difference (Final Values) = -1.8, 95% CI 2-sided [-7.9 to 4.2] — [estimate comment as in outcome 13, analysis 1]
Statistical Analysis 31: Comparison: Ipilimumab Plus gp100 vs gp100; Sleep disturbance change from baseline; Test type: Superiority or Other; p = 0.2450, ANCOVA; Mean Difference (Final Values) = -4.5, 95% CI 2-sided [-12.1 to 3.1] — [estimate comment as in outcome 13, analysis 1]
Statistical Analysis 32: Comparison: Ipilimumab Monotherapy vs gp100; Sleep disturbance change from baseline; Test type: Superiority or Other; p = 0.8464, ANCOVA; Mean Difference (Final Values) = -0.9, 95% CI 2-sided [-10.0 to 8.2] — [estimate comment as in outcome 13, analysis 1]
Statistical Analysis 33: Comparison: Ipilimumab Plus gp100 vs Ipilimumab Monotherapy; Sleep Disturbance change from baseline; Test type: Superiority or Other; p = 0.3351, ANCOVA; Mean Difference (Final Values) = -3.6, 95% CI 2-sided [-10.9 to 3.7] — [estimate comment as in outcome 13, analysis 1]
Statistical Analysis 34: Comparison: Ipilimumab Plus gp100 vs gp100; Appetite loss change from baseline; Test type: Superiority or Other; p = 0.6291, ANCOVA; Mean Difference (Final Values) = -1.8, 95% CI 2-sided [-9.1 to 5.5] — [estimate comment as in outcome 13, analysis 1]
Statistical Analysis 35: Comparison: Ipilimumab Monotherapy vs gp100; Appetite Loss change from baseline; Test type: Superiority or Other; p = 0.7675, ANCOVA; Mean Difference (Final Values) = 1.3, 95% CI 2-sided [-7.4 to 10.1] — [estimate comment as in outcome 13, analysis 1]
Statistical Analysis 36: Comparison: Ipilimumab Plus gp100 vs Ipilimumab Monotherapy; Appetite Loss change from baseline; Test type: Superiority or Other; p = 0.3911, ANCOVA; Mean Difference (Final Values) = -3.1, 95% CI 2-sided [-10.2 to 4.0] — [estimate comment as in outcome 13, analysis 1]
Statistical Analysis 37: Comparison: Ipilimumab Plus gp100 vs gp100; Constipation change from baseline; Test type: Superiority or Other; p = 0.0431, ANCOVA; Mean Difference (Final Values) = -6.5, 95% CI 2-sided [-12.9 to -0.2] — [estimate comment as in outcome 13, analysis 1]
Statistical Analysis 38: Comparison: Ipilimumab Monotherapy vs gp100; Constipation change from baseline; Test type: Superiority or Other; p = 0.0101, ANCOVA; Mean Difference (Final Values) = -9.9, 95% CI 2-sided [-17.4 to -2.4] — [estimate comment as in outcome 13, analysis 1]
Statistical Analysis 39: Comparison: Ipilimumab Plus gp100 vs Ipilimumab Monotherapy; Constipation change from baseline; Test type: Superiority or Other; p = 0.2796, ANCOVA; Mean Difference (Final Values) = 3.4, 95% CI 2-sided [-2.8 to 9.5] — [estimate comment as in outcome 13, analysis 1]
Statistical Analysis 40: Comparison: Ipilimumab Plus gp100 vs gp100; Diarrhea change from baseline; Test type: Superiority or Other; p = 0.1940, ANCOVA; Mean Difference (Final Values) = 4.3, 95% CI 2-sided [-2.2 to 10.8] — [estimate comment as in outcome 13, analysis 1]
Statistical Analysis 41: Comparison: Ipilimumab Monotherapy vs gp100; Diarrhea change from baseline; Test type: Superiority or Other; p = 0.0821, ANCOVA; Mean Difference (Final Values) = 6.9, 95% CI 2-sided [-0.9 to 14.8] — [estimate comment as in outcome 13, analysis 1]
Statistical Analysis 42: Comparison: Ipilimumab Plus gp100 vs Ipilimumab Monotherapy; Diarrhea change from baseline; Test type: Superiority or Other; p = 0.4169, ANCOVA; Mean Difference (Final Values) = -2.6, 95% CI 2-sided [-9.0 to 3.8] — [estimate comment as in outcome 13, analysis 1]
Statistical Analysis 43: Comparison: Ipilimumab Plus gp100 vs gp100; Financial Impact change from baseline; Test type: Superiority or Other; p = 0.5717, ANCOVA; Mean Difference (Final Values) = -1.7, 95% CI 2-sided [-7.5 to 4.2] — [estimate comment as in outcome 13, analysis 1]
Statistical Analysis 44: Comparison: Ipilimumab Monotherapy vs gp100; Financial Impact change from baseline; Test type: Superiority or Other; p = 0.6949, ANCOVA; Mean Difference (Final Values) = 1.4, 95% CI 2-sided [-5.6 to 8.4] — [estimate comment as in outcome 13, analysis 1]
Statistical Analysis 45: Comparison: Ipilimumab Plus gp100 vs Ipilimumab Monotherapy; Financial Impact change from baseline; Test type: Superiority or Other; p = 0.2849, ANCOVA; Mean Difference (Final Values) = -3.1, 95% CI 2-sided [-8.8 to 2.6] — [estimate comment as in outcome 13, analysis 1]

14. Secondary Outcome: Percentage of Participants With On-Study Adverse Events (AEs) and AEs With an Outcome of Death
Description: An AE was defined as any undesirable sign, symptom, clinically significant laboratory abnormality, or medical condition occurring after starting study treatment, even if the event was not considered to be treatment-related. Adverse events are graded using the Cancer Therapy Evaluation Program (CTEP) Common Terminology Criteria for Adverse Events (CTCAE), Version 3.0. If CTCAE grading does not exist for an adverse event, the intensity of mild (1), moderate (2), severe (3), and life-threatening (4) were used.
Time Frame: On-study adverse events include all AEs reported between the first dose and 70 days after the last dose of study therapy (end of the study was defined as the time at which 481 deaths were observed [264 weeks]).
Population: All subjects who received at least 1 dose or any partial dose of study medication.
Measure: Number; unit: percentage of participants
Arm/Group | Ipilimumab Plus gp100 | Ipilimumab Monotherapy | gp100
Number analyzed (Participants) | 380 | 131 | 132
percentage of participants
  Any On-Study AE | 98.4 | 96.9 | 97.0
  Severe (>=Grade 3) On-Study AEs | 50.8 | 55.0 | 52.3
  Serious On-Study AEs | 40.8 | 42.0 | 39.4
  Related On-Study AEs | 88.9 | 80.2 | 78.8
  On-Study AEs Leading to Discontinuation | 9.2 | 13.0 | 3.8
  AEs with Outcome of Death | 6.1 | 9.9 | 6.1
  Related AE with Outcome of Death | 2.1 | 3.1 | 1.5

15. Secondary Outcome: Percentage of Participants With Immune-Related Adverse Events (irAEs)
Description: An immune related adverse event (irAE) was defined as an adverse event of unknown etiology, associated with study drug exposure and consistent with an immune phenomenon. The irAEs were programmatically determined from a predefined list of MedDRA version 12.0 high-level group terms, high-level terms and preferred terms of all ipilimumab related adverse event. The category of "Other irAEs" includes blood, eye, immune, infections, renal, and respiratory systems.
Time Frame: as for outcome 14
Population: All subjects who received at least 1 dose or any partial dose of study medication.
Measure: Number; unit: percentage of participants
Arm/Group | Ipilimumab Plus gp100 | Ipilimumab Monotherapy | gp100
Number analyzed (Participants) | 380 | 131 | 132
percentage of participants
  Any On-Study irAEs | 58.2 | 61.1 | 31.8
  On-Study Severe irAEs | 11.3 | 15.3 | 3.0
  On-Study Serious irAEs | 10.5 | 13.0 | 0.8
  On-Study irAEs Leading to Discontinuation | 5.8 | 8.4 | 0.8
  Death Due to irAEs | 1.3 | 1.5 | 0
  Gastrointestinal irAEs (any grade) | 32.1 | 29.0 | 14.4
  Severe (>= Grade 3) Gastrointestinal irAEs | 6.3 | 7.6 | 0.8
  Liver irAEs (any grade) | 2.1 | 3.8 | 4.5
  Severe (>= Grade 3) Liver irAEs | 1.1 | 0.8 | 2.3
  Endocrine irAEs (any grade) | 3.9 | 7.6 | 1.5
  Severe (>= Grade 3) Endocrine irAEs | 1.1 | 3.8 | 0
  Skin irAEs (any grade) | 40.0 | 43.5 | 16.7
  Severe (>= Grade 3) Skin irAEs | 2.4 | 1.5 | 0
  Neurological irAEs (any grade) | 0.5 | 0 | 0
  Severe (>= Grade 3) Neurological irAEs | 0.5 | 0 | 0
  Other irAEs (any grade) | 3.2 | 4.6 | 2.3
  Severe (>= Grade 3) Other irAEs | 1.6 | 2.3 | 0.8

16. Secondary Outcome: Percentage of Participants With Worst On-Study Hematological Abnormalities
Description: ANC=Absolute Neutrophil Count. CTCAE v3.0 Grades 0 through 4 of severity for each AE based on this general guideline: Grade 0=Normal, Grade 1=Mild AE, Grade 2=Moderate AE, Grade 3=Severe AE, Grade 4=Life-threatening or disabling AE.
Time Frame: On-study laboratory results are results reported after the first dose date and within 70 days of last dose of study therapy (end of the study was defined as the time at which 481 deaths were observed [264 weeks]).
Population: All subjects who received at least 1 dose or any partial dose of study medication. N=Number of participants analyzed; n=number of participants with given laboratory evaluation.
Measure: Number; unit: percentage of participants
Arm/Group | Ipilimumab Plus gp100 | Ipilimumab Monotherapy | gp100
Number analyzed (Participants) | 380 | 131 | 132
percentage of participants
  Hemoglobin, Grade 0 (n=352, 121, 126) | 48.9 | 44.6 | 46.8
  Hemoglobin, Grade 1 (n=352, 121, 126) | 37.2 | 40.5 | 34.1
  Hemoglobin, Grade 2 (n=352, 121, 126) | 12.2 | 14.0 | 15.1
  Hemoglobin, Grade 3 (n=352, 121, 126) | 1.7 | 0.8 | 4.0
  Hemoglobin, Grade 4 (n=352, 121, 126) | 0 | 0 | 0
  Hemoglobin, Grade 1-4 (n=352, 121, 126) | 51.1 | 55.4 | 53.2
  Hemoglobin, Grade 3-4 (n=352, 121, 126) | 1.7 | 0.8 | 4.0
  White Blood Cells, Grade 0 (n=352, 121, 126) | 97.2 | 95.9 | 92.9
  White Blood Cells, Grade 1 (n=352, 121, 126) | 1.4 | 1.7 | 5.6
  White Blood Cells, Grade 2 (n=352, 121, 126) | 1.1 | 2.5 | 1.6
  White Blood Cells, Grade 3 (n=352, 121, 126) | 0.3 | 0 | 0
  White Blood Cells, Grade 4 (n=352, 121, 126) | 0 | 0 | 0
  White Blood Cells, Grade 1-4 (n=352, 121, 126) | 2.8 | 4.1 | 7.1
  White Blood Cells, Grade 3-4 (n=352, 121, 126) | 0.3 | 0 | 0
  ANC, Grade 0 (n=352, 121, 126) | 95.5 | 93.4 | 96.0
  ANC, Grade 1 (n=352, 121, 126) | 2.8 | 3.3 | 2.4
  ANC, Grade 2 (n=352, 121, 126) | 0.9 | 2.5 | 0.8
  ANC, Grade 3 (n=352, 121, 126) | 0.6 | 0.8 | 0.8
  ANC, Grade 4 (n=352, 121, 126) | 0.3 | 0 | 0
  ANC, Grade 1-4 (n=352, 121, 126) | 4.5 | 6.6 | 4.0
  ANC, Grade 3-4 (n=352, 121, 126) | 0.9 | 0.8 | 0.8
  Platelet Count, Grade 0 (n=349, 121, 126) | 94.6 | 90.1 | 91.3
  Platelet Count, Grade 1 (n=349, 121, 126) | 4.9 | 9.1 | 8.7
  Platelet Count, Grade 2 (n=349, 121, 126) | 0.6 | 0.8 | 0
  Platelet Count, Grade 3 (n=349, 121, 126) | 0 | 0 | 0
  Platelet Count, Grade 4 (n=349, 121, 126) | 0 | 0 | 0
  Platelet Count, Grade 1-4 (n=349, 121, 126) | 5.4 | 9.9 | 8.7
  Platelet Count, Grade 3-4 (n=349, 121, 126) | 0 | 0 | 0
  Lymphocytes (absolute), Grade 0 (n=352, 121, 126) | 33.8 | 34.7 | 22.2
  Lymphocytes (absolute), Grade 1 (n=352, 121, 126) | 46.3 | 47.9 | 42.9
  Lymphocytes (absolute), Grade 2 (n=352, 121, 126) | 15.1 | 14.9 | 25.4
  Lymphocytes (absolute), Grade 3 (n=352, 121, 126) | 4.3 | 2.5 | 9.5
  Lymphocytes (absolute), Grade 4 (n=352, 121, 126) | 0.6 | 0 | 0
  Lymphocytes (absolute), Grade 1-4(n=352, 121, 126) | 66.2 | 65.3 | 77.8
  Lymphocytes (absolute), Grade 3-4(n=352, 121, 126) | 4.8 | 2.5 | 9.5

17. Secondary Outcome: Percentage of Participants With Worst On-Study Liver Abnormalities
Description: ALT=alanine aminotransferase; AST=aspartate aminotransferase. CTCAE v3.0 Grades 0 through 4 of severity for each AE based on this general guideline: Grade 0=Normal, Grade 1=Mild AE, Grade 2=Moderate AE, Grade 3=Severe AE, Grade 4=Life-threatening or disabling AE.
Time Frame: as for outcome 14
Population: as for outcome 16
Measure: Number; unit: percentage of participants
Arm/Group | Ipilimumab Plus gp100 | Ipilimumab Monotherapy | gp100
Number analyzed (Participants) | 380 | 131 | 132
percentage of participants
  ALT, Grade 0 (n=352, 121, 126) | 83.2 | 76.0 | 84.9
  ALT, Grade 1 (n=352, 121, 126) | 13.6 | 19.0 | 12.7
  ALT, Grade 2 (n=352, 121, 126) | 2.0 | 3.3 | 1.6
  ALT, Grade 3 (n=352, 121, 126) | 0.9 | 1.7 | 0.8
  ALT, Grade 4 (n=352, 121, 126) | 0.3 | 0 | 0
  ALT, Grade 1-4 (n=352, 121, 126) | 16.8 | 24.0 | 15.1
  ALT, Grade 3-4 (n=352, 121, 126) | 1.1 | 1.7 | 0.8
  AST, Grade 0 (n=352, 121, 126) | 80.4 | 71.9 | 81.7
  AST, Grade 1 (n=352, 121, 126) | 16.5 | 23.1 | 15.1
  AST, Grade 2 (n=352, 121, 126) | 1.4 | 3.3 | 2.4
  AST, Grade 3 (n=352, 121, 126) | 1.4 | 1.7 | 0.8
  AST, Grade 4 (n=352, 121, 126) | 0.3 | 0 | 0
  AST, Grade 1-4 (n=352, 121, 126) | 19.6 | 28.1 | 18.3
  AST, Grade 3-4 (n=352, 121, 126) | 1.7 | 1.7 | 0.8
  Total Bilirubin, Grade 0 (n=353, 121, 127) | 95.5 | 93.4 | 98.4
  Total Bilirubin, Grade 1 (n=353, 121, 127) | 2.5 | 4.1 | 0.8
  Total Bilirubin, Grade 2 (n=353, 121, 127) | 1.4 | 1.7 | 0.8
  Total Bilirubin, Grade 3 (n=353, 121, 127) | 0.6 | 0.8 | 0
  Total Bilirubin, Grade 4 (n=353, 121, 127) | 0 | 0 | 0
  Total Bilirubin, Grade 1-4 (n=353, 121, 127) | 4.5 | 6.6 | 1.6
  Total Bilirubin, Grade 3-4 (n=353, 121, 127) | 0.6 | 0.8 | 0
  Alkaline Phosphatase, Grade 0 (n=353, 121, 128) | 73.7 | 71.9 | 71.1
  Alkaline Phosphatase, Grade 1 (n=353, 121, 128) | 19.8 | 20.7 | 24.2
  Alkaline Phosphatase, Grade 2 (n=353, 121, 128) | 4.8 | 4.1 | 3.9
  Alkaline Phosphatase, Grade 3 (n=353, 121, 128) | 1.7 | 3.3 | 0.8
  Alkaline Phosphatase, Grade 4 (n=353, 121, 128) | 0 | 0 | 0
  Alkaline Phosphatase, Grade 1-4 (n=353, 121, 128) | 26.3 | 28.1 | 28.9
  Alkaline Phosphatase, Grade 3-4 (n=353, 121, 128) | 1.7 | 3.3 | 0.8

18. Secondary Outcome: Percentage of Participants With Worst On-Study Renal Abnormalities
Description: CTCAE v3.0 Grades 0 through 4 of severity for each AE based on this general guideline: Grade 0=Normal, Grade 1=Mild AE, Grade 2=Moderate AE, Grade 3=Severe AE, Grade 4=Life-threatening or disabling AE.
Time Frame: as for outcome 14
Population: as for outcome 16
Measure: Number; unit: percentage of participants
Arm/Group | Ipilimumab Plus gp100 | Ipilimumab Monotherapy | gp100
Number analyzed (Participants) | 380 | 131 | 132
percentage of participants
  Creatinine, Grade 0 (n=353, 121, 128) | 89.5 | 88.4 | 88.3
  Creatinine, Grade 1 (n=353, 121, 128) | 8.8 | 9.9 | 9.4
  Creatinine, Grade 2 (n=353, 121, 128) | 1.4 | 1.7 | 2.3
  Creatinine, Grade 3 (n=353, 121, 128) | 0.3 | 0 | 0
  Creatinine, Grade 4 (n=353, 121, 128) | 0 | 0 | 0
  Creatinine, Grade 1-4 (n=353, 121, 128) | 10.5 | 11.6 | 11.7
  Creatinine, Grade 3-4 (n=353, 121, 128) | 0.3 | 0 | 0

19. Secondary Outcome: Clinically Meaningful Changes in Vital Signs and Physical Examinations
Description: Clinically meaningful changes were according to investigator. Vital sign measurements include height, weight, temperature, pulse, and resting systolic and diastolic blood pressure.
Time Frame: vital signs and physical examination were evaluated at screening and at Weeks 1, 4, 7, 10, 12, 16, 20, 24, 28, 36, and every 3 months thereafter
Population: All subjects who received at least 1 dose or any partial dose of study medication.
Measure: Number; unit: participants
Arm/Group | Ipilimumab Plus gp100 | Ipilimumab Monotherapy | gp100
Number analyzed (Participants) | 380 | 131 | 132
participants
  Clinically Meaningful Vital Sign Changes | 0 | 0 | 0
  Clinically Meaningful Physical Examination Changes | 0 | 0 | 0

ADVERSE EVENTS:
Arm/Group | Ipilimumab Monotherapy | Ipilimumab Plus gp100 | gp100
Serious Adverse Events (participants affected / at risk) | 55/131 | 155/380 | 52/132
Other Adverse Events (participants affected / at risk) | 124/131 | 362/380 | 124/132
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ipilimumab Monotherapy (N=131) | Ipilimumab Plus gp100 (N=380) | gp100 (N=132)
ABDOMINAL DISTENSION (Gastrointestinal disorders) | 1 | 1 | 0
ABDOMINAL PAIN (Gastrointestinal disorders) | 2 | 4 | 5
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 0 | 2 | 0
ABDOMINAL WALL MASS (Gastrointestinal disorders) | 0 | 1 | 0
ACCIDENTAL OVERDOSE (Injury, poisoning and procedural complications) | 0 | 1 | 0
ACUTE HEPATIC FAILURE (Hepatobiliary disorders) | 1 | 0 | 0
ACUTE PULMONARY OEDEMA (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
ACUTE RESPIRATORY DISTRESS SYNDROME (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
ADRENAL INSUFFICIENCY (Endocrine disorders) | 1 | 1 | 0
ADVERSE EVENT (General disorders) | 1 | 3 | 0
ANAEMIA (Blood and lymphatic system disorders) | 4 | 5 | 5
ANGIOPATHY (Vascular disorders) | 1 | 0 | 0
ANXIETY (Psychiatric disorders) | 0 | 0 | 1
APHASIA (Nervous system disorders) | 0 | 1 | 0
APPENDICITIS (Infections and infestations) | 0 | 1 | 0
ARTERIAL THROMBOSIS LIMB (Vascular disorders) | 1 | 0 | 0
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
ASCITES (Gastrointestinal disorders) | 1 | 1 | 0
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 0 | 0 | 1
ASTHENIA (General disorders) | 3 | 4 | 1
ATAXIA (Nervous system disorders) | 0 | 0 | 1
ATONIC URINARY BLADDER (Renal and urinary disorders) | 0 | 1 | 0
ATRIAL FIBRILLATION (Cardiac disorders) | 0 | 1 | 1
BACK PAIN (Musculoskeletal and connective tissue disorders) | 0 | 2 | 2
BACTERAEMIA (Infections and infestations) | 0 | 1 | 0
BASAL CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
BILE DUCT OBSTRUCTION (Hepatobiliary disorders) | 0 | 1 | 0
BLADDER PAIN (Renal and urinary disorders) | 0 | 1 | 0
BLOOD CORTICOTROPHIN DECREASED (Investigations) | 1 | 0 | 0
BONE PAIN (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
BRAIN OEDEMA (Nervous system disorders) | 1 | 2 | 0
BREAST MASS (Reproductive system and breast disorders) | 0 | 0 | 1
BRONCHIAL OBSTRUCTION (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
BRONCHOPNEUMONIA (Infections and infestations) | 1 | 1 | 0
CANCER PAIN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
CARDIAC FAILURE (Cardiac disorders) | 1 | 1 | 0
CARDIAC FAILURE CONGESTIVE (Cardiac disorders) | 1 | 1 | 0
CARDIAC TAMPONADE (Cardiac disorders) | 0 | 1 | 0
CARDIOPULMONARY FAILURE (Cardiac disorders) | 0 | 1 | 0
CATHETER RELATED INFECTION (Infections and infestations) | 0 | 1 | 0
CELLULITIS (Infections and infestations) | 0 | 1 | 1
CEREBRAL HAEMORRHAGE (Nervous system disorders) | 0 | 0 | 2
CEREBROVASCULAR ACCIDENT (Nervous system disorders) | 0 | 1 | 0
CHEST PAIN (General disorders) | 0 | 0 | 1
CHILLS (General disorders) | 0 | 1 | 0
CHOLECYSTITIS (Hepatobiliary disorders) | 1 | 0 | 0
COLITIS (Gastrointestinal disorders) | 7 | 14 | 0
COMA (Nervous system disorders) | 0 | 1 | 1
CONFUSIONAL STATE (Psychiatric disorders) | 2 | 1 | 1
CONSTIPATION (Gastrointestinal disorders) | 0 | 3 | 1
CONVULSION (Nervous system disorders) | 0 | 1 | 1
CORONARY ARTERY DISEASE (Cardiac disorders) | 1 | 0 | 0
COUGH (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
CYSTITIS (Infections and infestations) | 0 | 1 | 0
DECREASED APPETITE (Metabolism and nutrition disorders) | 2 | 3 | 1
DEEP VEIN THROMBOSIS (Vascular disorders) | 2 | 5 | 1
DEHYDRATION (Metabolism and nutrition disorders) | 1 | 8 | 4
DELIRIUM (Psychiatric disorders) | 0 | 1 | 0
DEPRESSED LEVEL OF CONSCIOUSNESS (Nervous system disorders) | 0 | 1 | 0
DIARRHOEA (Gastrointestinal disorders) | 6 | 16 | 0
DISEASE PROGRESSION (General disorders) | 2 | 6 | 3
DIZZINESS (Nervous system disorders) | 0 | 0 | 2
DYSARTHRIA (Nervous system disorders) | 0 | 1 | 0
DYSPHAGIA (Gastrointestinal disorders) | 1 | 0 | 1
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 3 | 2 | 7
ENTEROCOCCAL BACTERAEMIA (Infections and infestations) | 1 | 0 | 0
EPIDURITIS (Nervous system disorders) | 0 | 0 | 1
ERYSIPELAS (Infections and infestations) | 0 | 0 | 1
EYELID INFECTION (Infections and infestations) | 0 | 1 | 0
FAILURE TO THRIVE (Metabolism and nutrition disorders) | 0 | 2 | 0
FATIGUE (General disorders) | 1 | 0 | 0
FEMORAL NECK FRACTURE (Injury, poisoning and procedural complications) | 0 | 0 | 1
GAIT DISTURBANCE (General disorders) | 1 | 0 | 1
GAMMA-GLUTAMYLTRANSFERASE INCREASED (Investigations) | 0 | 0 | 1
GASTRITIS (Gastrointestinal disorders) | 0 | 2 | 0
GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 0 | 2 | 0
GASTROINTESTINAL INFECTION (Infections and infestations) | 0 | 1 | 0
GASTROINTESTINAL PERFORATION (Gastrointestinal disorders) | 0 | 1 | 0
GASTROINTESTINAL STOMA COMPLICATION (Injury, poisoning and procedural complications) | 0 | 1 | 0
GENERAL PHYSICAL HEALTH DETERIORATION (General disorders) | 0 | 2 | 2
GENERALISED OEDEMA (General disorders) | 1 | 0 | 0
GLOMERULONEPHRITIS (Renal and urinary disorders) | 1 | 0 | 0
GUILLAIN-BARRE SYNDROME (Nervous system disorders) | 0 | 1 | 0
HAEMATOCHEZIA (Gastrointestinal disorders) | 0 | 2 | 0
HAEMATOMA (Vascular disorders) | 0 | 1 | 1
HAEMOLYTIC ANAEMIA (Blood and lymphatic system disorders) | 0 | 1 | 0
HAEMOPTYSIS (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
HAEMORRHAGE INTRACRANIAL (Nervous system disorders) | 0 | 2 | 0
HAEMORRHOIDS (Gastrointestinal disorders) | 0 | 1 | 0
HAEMOTHORAX (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
HEADACHE (Nervous system disorders) | 0 | 2 | 1
HEPATIC FAILURE (Hepatobiliary disorders) | 1 | 1 | 0
HEPATITIS (Hepatobiliary disorders) | 0 | 1 | 0
HEPATITIS A (Infections and infestations) | 1 | 0 | 0
HEPATITIS B (Infections and infestations) | 1 | 0 | 0
HERNIA OBSTRUCTIVE (General disorders) | 0 | 1 | 0
HIP FRACTURE (Injury, poisoning and procedural complications) | 0 | 1 | 0
HYDROCEPHALUS (Nervous system disorders) | 0 | 1 | 0
HYDRONEPHROSIS (Renal and urinary disorders) | 0 | 1 | 0
HYPERBILIRUBINAEMIA (Hepatobiliary disorders) | 0 | 1 | 0
HYPERTENSIVE CRISIS (Vascular disorders) | 0 | 0 | 1
HYPOAESTHESIA (Nervous system disorders) | 0 | 1 | 0
HYPOALBUMINAEMIA (Metabolism and nutrition disorders) | 1 | 0 | 0
HYPOGLYCAEMIA (Metabolism and nutrition disorders) | 1 | 0 | 0
HYPOGONADISM (Endocrine disorders) | 0 | 1 | 0
HYPONATRAEMIA (Metabolism and nutrition disorders) | 0 | 1 | 0
HYPOPHAGIA (Metabolism and nutrition disorders) | 0 | 1 | 0
HYPOPHYSITIS (Endocrine disorders) | 2 | 1 | 0
HYPOPITUITARISM (Endocrine disorders) | 2 | 3 | 0
HYPOTENSION (Vascular disorders) | 3 | 1 | 2
HYPOTHYROIDISM (Endocrine disorders) | 0 | 1 | 0
ILEUS (Gastrointestinal disorders) | 0 | 3 | 0
INFECTION (Infections and infestations) | 1 | 1 | 0
INFLUENZA LIKE ILLNESS (General disorders) | 1 | 0 | 0
INFUSION RELATED REACTION (General disorders) | 0 | 1 | 0
INJECTION SITE REACTION (General disorders) | 0 | 1 | 0
INJECTION SITE ULCER (General disorders) | 0 | 1 | 0
INTERNATIONAL NORMALISED RATIO ABNORMAL (Investigations) | 0 | 1 | 0
INTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 0 | 1 | 0
INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 0 | 2 | 0
INTESTINAL PERFORATION (Gastrointestinal disorders) | 0 | 3 | 0
INTRACRANIAL PRESSURE INCREASED (Nervous system disorders) | 0 | 1 | 0
INTRACRANIAL TUMOUR HAEMORRHAGE (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
INTUSSUSCEPTION (Gastrointestinal disorders) | 0 | 0 | 2
IRIDOCYCLITIS (Eye disorders) | 0 | 1 | 0
JAUNDICE (Hepatobiliary disorders) | 0 | 1 | 0
JAUNDICE CHOLESTATIC (Hepatobiliary disorders) | 0 | 1 | 0
LARGE INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 1 | 0 | 0
LARGE INTESTINE PERFORATION (Gastrointestinal disorders) | 0 | 2 | 0
LETHARGY (Nervous system disorders) | 0 | 2 | 0
LEUKOCYTOCLASTIC VASCULITIS (Skin and subcutaneous tissue disorders) | 0 | 2 | 0
LEUKOCYTOSIS (Blood and lymphatic system disorders) | 0 | 1 | 0
LOCALISED INFECTION (Infections and infestations) | 1 | 0 | 0
LOWER RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 | 1 | 0
LYMPHOEDEMA (Vascular disorders) | 0 | 0 | 1
MALIGNANT ASCITES (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
MALIGNANT MELANOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 3 | 1
MALIGNANT NEOPLASM PROGRESSION (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 3 | 0
MALNUTRITION (Metabolism and nutrition disorders) | 0 | 1 | 0
MENINGEAL DISORDER (Nervous system disorders) | 0 | 2 | 0
MENINGITIS (Infections and infestations) | 0 | 1 | 0
MENTAL STATUS CHANGES (Psychiatric disorders) | 0 | 2 | 0
METASTASES TO BREAST (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
METASTASES TO CENTRAL NERVOUS SYSTEM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 3 | 0
METASTASES TO SPINE (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
METASTATIC MALIGNANT MELANOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
METASTATIC NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
METASTATIC PAIN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 3 | 0
MULTI-ORGAN FAILURE (General disorders) | 0 | 2 | 2
MUSCULAR WEAKNESS (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0
MYOCLONUS (Nervous system disorders) | 1 | 0 | 0
NAUSEA (Gastrointestinal disorders) | 2 | 6 | 4
NECK PAIN (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
NEUTROPENIA (Blood and lymphatic system disorders) | 1 | 1 | 0
OEDEMA (General disorders) | 2 | 1 | 0
OEDEMA PERIPHERAL (General disorders) | 1 | 1 | 0
PAIN (General disorders) | 1 | 3 | 0
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 0 | 3 | 1
PAINFUL RESPIRATION (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
PATHOLOGICAL FRACTURE (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
PELVIC PAIN (Reproductive system and breast disorders) | 0 | 1 | 0
PERICARDIAL EFFUSION (Cardiac disorders) | 0 | 1 | 0
PERIRECTAL ABSCESS (Infections and infestations) | 1 | 0 | 0
PERITONITIS (Gastrointestinal disorders) | 0 | 1 | 0
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 2 | 5 | 4
PLEURITIC PAIN (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
PNEUMONIA (Infections and infestations) | 2 | 8 | 3
PNEUMONITIS (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
POLYMYALGIA RHEUMATICA (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
POSTOPERATIVE WOUND INFECTION (Infections and infestations) | 0 | 1 | 0
PROCEDURAL COMPLICATION (Injury, poisoning and procedural complications) | 0 | 1 | 0
PROCTALGIA (Gastrointestinal disorders) | 1 | 0 | 0
PSEUDOMONAL SEPSIS (Infections and infestations) | 0 | 1 | 0
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 2
PULMONARY HAEMORRHAGE (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
PYREXIA (General disorders) | 2 | 7 | 1
RASH (Skin and subcutaneous tissue disorders) | 0 | 2 | 0
RASH GENERALISED (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
RASH PRURITIC (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
RECTAL STENOSIS (Gastrointestinal disorders) | 0 | 1 | 0
RENAL FAILURE (Renal and urinary disorders) | 3 | 3 | 0
RENAL FAILURE ACUTE (Renal and urinary disorders) | 0 | 0 | 1
RENAL TUBULAR NECROSIS (Renal and urinary disorders) | 0 | 1 | 0
RESPIRATORY ARREST (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
RESPIRATORY DEPRESSION (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 0
SEPSIS (Infections and infestations) | 3 | 4 | 0
SEPTIC SHOCK (Infections and infestations) | 1 | 1 | 1
SLEEP APNOEA SYNDROME (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
SMALL INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 0 | 0 | 1
SPINAL CORD COMPRESSION (Nervous system disorders) | 1 | 3 | 0
SUPERIOR VENA CAVAL OCCLUSION (Vascular disorders) | 0 | 1 | 0
SUPRAVENTRICULAR TACHYCARDIA (Cardiac disorders) | 1 | 0 | 0
SYNCOPE (Nervous system disorders) | 1 | 1 | 0
TACHYCARDIA (Cardiac disorders) | 0 | 1 | 0
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 1 | 0 | 0
THROMBOSIS (Vascular disorders) | 1 | 1 | 0
TOXIC EPIDERMAL NECROLYSIS (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
TUMOUR HAEMORRHAGE (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 2
TUMOUR LYSIS SYNDROME (Metabolism and nutrition disorders) | 1 | 0 | 0
TUMOUR PAIN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 2 | 1
UPPER GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 0 | 1 | 0
URETERIC OBSTRUCTION (Renal and urinary disorders) | 0 | 1 | 0
URINARY INCONTINENCE (Renal and urinary disorders) | 0 | 1 | 1
URINARY RETENTION (Renal and urinary disorders) | 0 | 2 | 0
URINARY TRACT INFECTION (Infections and infestations) | 0 | 2 | 3
URINE OUTPUT DECREASED (Investigations) | 1 | 0 | 0
VOMITING (Gastrointestinal disorders) | 3 | 7 | 3
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ipilimumab Monotherapy (N=131) | Ipilimumab Plus gp100 (N=380) | gp100 (N=132)
ABDOMINAL DISTENSION (Gastrointestinal disorders) | 0 | 13 | 9
ABDOMINAL PAIN (Gastrointestinal disorders) | 20 | 64 | 18
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 7 | 17 | 11
ADVERSE EVENT (General disorders) | 4 | 22 | 5
ANAEMIA (Blood and lymphatic system disorders) | 14 | 36 | 22
ANXIETY (Psychiatric disorders) | 5 | 31 | 9
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 12 | 30 | 14
ASTHENIA (General disorders) | 6 | 37 | 17
BACK PAIN (Musculoskeletal and connective tissue disorders) | 9 | 32 | 16
CHILLS (General disorders) | 9 | 23 | 7
CONSTIPATION (Gastrointestinal disorders) | 27 | 79 | 34
COUGH (Respiratory, thoracic and mediastinal disorders) | 21 | 55 | 17
DECREASED APPETITE (Metabolism and nutrition disorders) | 33 | 85 | 29
DIARRHOEA (Gastrointestinal disorders) | 41 | 142 | 26
DIZZINESS (Nervous system disorders) | 5 | 27 | 13
DYSPEPSIA (Gastrointestinal disorders) | 2 | 14 | 10
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 16 | 45 | 20
ERYTHEMA (Skin and subcutaneous tissue disorders) | 10 | 26 | 7
FATIGUE (General disorders) | 55 | 137 | 41
FLATULENCE (Gastrointestinal disorders) | 3 | 9 | 8
HEADACHE (Nervous system disorders) | 19 | 64 | 18
HOT FLUSH (Vascular disorders) | 6 | 8 | 8
HYPERHIDROSIS (Skin and subcutaneous tissue disorders) | 6 | 14 | 12
HYPOTENSION (Vascular disorders) | 8 | 12 | 4
INFLUENZA LIKE ILLNESS (General disorders) | 7 | 20 | 3
INJECTION SITE ERYTHEMA (General disorders) | 1 | 26 | 5
INJECTION SITE INDURATION (General disorders) | 0 | 25 | 4
INJECTION SITE PAIN (General disorders) | 2 | 25 | 13
INJECTION SITE REACTION (General disorders) | 2 | 109 | 26
INSOMNIA (Psychiatric disorders) | 16 | 33 | 15
MUSCULOSKELETAL CHEST PAIN (Musculoskeletal and connective tissue disorders) | 7 | 7 | 2
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 5 | 30 | 10
MYALGIA (Musculoskeletal and connective tissue disorders) | 8 | 28 | 4
NAUSEA (Gastrointestinal disorders) | 44 | 127 | 49
OEDEMA PERIPHERAL (General disorders) | 12 | 47 | 22
PAIN (General disorders) | 6 | 23 | 15
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 9 | 51 | 19
PRURITUS (Skin and subcutaneous tissue disorders) | 39 | 79 | 14
PYREXIA (General disorders) | 15 | 74 | 23
RASH (Skin and subcutaneous tissue disorders) | 29 | 78 | 9
URINARY TRACT INFECTION (Infections and infestations) | 8 | 8 | 4
VOMITING (Gastrointestinal disorders) | 30 | 71 | 27
WEIGHT DECREASED (Investigations) | 8 | 33 | 12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.